CLINICAL TRIAL: NCT06041672
Title: The Effectiveness of Warm Hand Bath in Improving Anxiety Before Lower Limbs Surgery Among Middle-aged and Older Patients
Brief Title: The Effectiveness of Warm Hand Bath in Improving Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cathay General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CGH-P112023
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-08

CONDITIONS: Preoperative Anxiety
Keywords: lower limb bone surgery; warm water hand bath; preoperative anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Water Hand Baths (Experimental): Patients in the experimental group have their hand immersed in warm water (40°C) for ten minutes.
  Interventions: Behavioral: Warm Water Hand Baths
- Routine care (No Intervention): Including preoperative instructions, postoperative care, and monitoring of vital signs.

INTERVENTIONS:
Behavioral: Warm Water Hand Baths — 1. Patients in the experimental group receive warm water hand baths as an intervention on the evening before surgery.
  2. The intervention is carried out in the patient's room, room temperature was adjusted to 26°C and the timing is determined based on the patient's preference.
  3. The study utilizes a foldable water bucket with temperature maintenance capability.Patients in the experimental group have their hand immersed in warm water (40°C) for ten minutes in a comfortable lying position.
  Arms: Warm Water Hand Baths

SUMMARY:
Patients undergoing surgery often experience anxiety before the procedure. The aim of this study is to investigate the effectiveness of warm water baths in reducing preoperative anxiety levels in middle-aged and elderly patients undergoing lower limb orthopedic surgery. This study utilizes a randomized controlled trial design and focuses on middle-aged and elderly patients undergoing lower limb orthopedic surgery in the orthopedic ward of a medical center in northern Taiwan. The patients are divided into an experimental group and a control group using block randomization. Patients in the experimental group receive a 10-minute warm water bath at 40°C on the evening before surgery as an intervention, while the control group receives standard care. Data are collected from both groups before and after the intervention, including personal information, the State-Trait Anxiety Inventory, Visual Analog Scale for pain assessment, and Visual Analog Scale for relaxation, as well as vital sign measurements. Statistical analysis of the data is conducted using SPSS version 18.0 software, employing mean values, standard deviations, percentages, independent t-tests, chi-square tests, paired-sample t-tests, and generalized estimating equations for data analysis.

DETAILED DESCRIPTION:
As the world's population ages, musculoskeletal surgeries have become a primary reason for surgery in elderly individuals, affecting 41.3% of elderly patients. Hospitalization and surgery can cause anxiety, and previous research has shown that the prevalence of preoperative anxiety in surgical patients is around 60-94%, with over 35% of cases experiencing high levels of anxiety. When patients experience preoperative anxiety, it can affect their postoperative recovery, including wound healing, functional recovery, the occurrence of complications, and increased length of hospital stay or recovery time. Early intervention to help patients relieve anxiety can reduce these negative effects. Current literature has shown that multimedia educational health education, music therapy, aromatherapy, massage, and other interventions can effectively reduce preoperative anxiety, but these interventions require professional training or the preparation of additional materials and equipment. In this study, a warm water hand bath was used as the intervention, mainly because lower limb surgery patients are not suitable for foot baths to achieve relaxation, and the operation of hand baths is simple, the equipment (warm water and basin) is easy to obtain, and patients or family members can easily learn to use it, making it convenient and accessible.Therefore, this study aims to understand how middle-aged and elderly participants who are about to undergo lower limb surgery can improve their preoperative anxiety, pain, and relaxation through the intervention of warm water hand baths.

After obtaining approval from the Taipei Cathay General Hospital Human Research Ethics Committee and registering on ClinicalTrials.gov, and obtaining consent from the Cathay Surgical Ward, the recruitment process began.

1. On the day of admission, subjects were recruited. Researcher (Principal Investigator ) personally introduced the study's purpose, recruitment procedure, and rights and obligations to eligible subjects. If the subjects expressed their willingness to participate, they were asked to sign an informed consent form.
2. Researcher used the admission time of the subjects as the recruitment time point. According to the order of subjects' admission, they were sequentially assigned to either the experimental group or the control group. An individual not involved in the study used a computer software program to generate serial numbers for randomization in blocks. The serial numbers and group assignments were placed in opaque envelopes with consecutive codes. After obtaining informed consent from the subjects, the envelopes were opened in sequence, and participants were assigned to the control or experimental group until a total of 78 subjects were recruited.
3. After knowing the subjects' group assignments, Researcher discussed the intervention time with the subjects. It was scheduled for the evening before the surgery, and subjects could choose a suitable time. The intervention took place in the subjects' hospital rooms.
4. Ten minutes before the warm water hand bath intervention, Researcher used the Braun ThermoScan® PRO 6000 ear thermometer and Omron HBP-1300 blood pressure monitor to measure vital signs (temperature, blood pressure, heart rate, respiration) and collected baseline questionnaire data. Questionnaires were administered on paper, and assistance was provided if subjects were unable to fill them out independently.
5. This study employed a foldable water bucket with temperature maintenance functionality for warm water hand baths. The water bucket did not require electricity but could maintain water temperature without it rising. Testing indicated that at room temperature (26°C), it could maintain water temperature for approximately 10 minutes. Subjects received the warm water hand bath the night before surgery, with the room temperature set at 26°C. If the subject's hospital room was not a single-person room, Researcher A negotiated the room temperature with adjacent patients. Four liters of 40°C warm water were added to the temperature-maintaining water bucket. To ensure temperature control, a floating LED water temperature monitor was used continuously. The monitor was the Dr.AV Saint Gok Technology-GE-53C Multi-Purpose Electronic Thermometer. If there was a drop in water temperature during the intervention, additional warm water was added to maintain the appropriate temperature. Due to potential pain and difficulty sitting up, subjects assumed a comfortable lying position with a blanket placed under their arm. The temperature-maintaining water bucket was placed on both sides of the bed, and Researcher A assisted the subjects in placing their hand into the water. The entire hand was immersed up to the wrist crease, approximately 5 centimeters, and soaked for ten minutes. After each use, subjects rinsed their hand thoroughly with clean water, followed by disinfection with 75% alcohol. After ensuring dryness, the equipment was stored to prevent potential alcohol-related hazards. The control group's room temperature was also adjusted to 26°C. Subjects assumed a comfortable lying position and received routine care, including preoperative instructions, postoperative care, and monitoring of vital signs.
6. Researcher conducted post-intervention measurements of vital signs (temperature, blood pressure, heart rate, respiration) and collected post-test questionnaire data for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age must be forty-five years or older.
2. Individuals diagnosed by a physician with lower limb bone-related conditions and planning to undergo orthopedic surgery.
3. Must maintain clear consciousness and be able to communicate verbally.
4. Patients with heart disease or diabetes must seek the opinion of the attending physicians (Dr. Liu Zhe-wei and Dr. Chen Yi-zhi) before undergoing this intervention.
5. The study encompasses the following lower limb orthopedic surgeries:

Total joint replacement surgery, including knee and hip joint replacements. Revision surgery for joint replacements. Joint osteotomy correction surgery. Arthroscopic joint surgery. Open reduction and internal fixation surgery. Other surgeries related to lower limb musculoskeletal conditions.

Exclusion Criteria:

1. Patients with hand or wrist fractures.
2. Individuals with peripheral circulation abnormalities.
3. Patients with autonomic nervous system disorders who are taking anxiety-related medications.
4. Pregnant women.
5. Individuals with wounds, infections, swelling, or injuries on the skin of both palms, preventing immersion in water.
6. Those suffering from other major illnesses or scheduled for two or more surgeries.
7. Patients requiring physiological monitoring.
8. Individuals needing a catheter placed below the wrist.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory,A-State,STAI-S | Baseline, before the intervention(T0)
  The questionnaire consists of 20 items, and research subjects are asked to select the response that best represents their current feelings of anxiety for each item. It is scored on a four-point Likert scale, with responses ranging from "Not at all" (scored as 1 point), "Somewhat" (scored as 2 points), "Moderately so" (scored as 3 points), to "Very much so" (scored as 4 points). Among the 20 items, 10 are reverse-scored (items 3, 4, 6, 7, 9, 12, 13, 14, 17, and 18), meaning that the scoring is reversed for these items. The total score ranges from 20 to 80 points, with higher scores indicating a higher level of anxiety.
State-Trait Anxiety Inventory,A-State,STAI-S | Immediately following after the intervention(T1)
  The questionnaire consists of 20 items, and research subjects are asked to select the response that best represents their current feelings of anxiety for each item. It is scored on a four-point Likert scale, with responses ranging from "Not at all" (scored as 1 point), "Somewhat" (scored as 2 points), "Moderately so" (scored as 3 points), to "Very much so" (scored as 4 points). Among the 20 items, 10 are reverse-scored (items 3, 4, 6, 7, 9, 12, 13, 14, 17, and 18), meaning that the scoring is reversed for these items. The total score ranges from 20 to 80 points, with higher scores indicating a higher level of anxiety.

SECONDARY OUTCOMES:
The pain(Visual Analogue Scale, VAS) | Baseline, before the intervention(T0)
  This type of pain assessment tool is commonly known as a visual analogue scale (VAS) and is used to quantify the subjective experience of pain by having individuals mark their level of pain on the line.
  A horizontal line that is 10 centimeters long is used to assess pain intensity. On this line, 0 centimeters on the left side represents "no pain," while 10 centimeters on the right side represents "extremely severe pain." Higher scores on this line indicate a higher level of pain intensity.
The pain(Visual Analogue Scale, VAS) | Immediately following after the intervention(T1)
  This type of pain assessment tool is commonly known as a visual analogue scale (VAS) and is used to quantify the subjective experience of pain by having individuals mark their level of pain on the line.
  A horizontal line that is 10 centimeters long is used to assess pain intensity. On this line, 0 centimeters on the left side represents "no pain," while 10 centimeters on the right side represents "extremely severe pain." Higher scores on this line indicate a higher level of pain intensity.
The Relaxation (Visual Analogue Scale,VAS) | Baseline, before the intervention(T0)
  The Relaxation VAS uses a continuous horizontal line that is 10 centimeters long. On this line, 0 centimeters on the left side represents "unable to relax," while 10 centimeters on the right side represents "extremely relaxed." The closer the mark is to 10 centimeters, the higher the level of relaxation. This scale allows individuals to subjectively indicate their degree of relaxation by marking a point on the line.
The Relaxation (Visual Analogue Scale,VAS) | Immediately following after the intervention(T1)
  The Relaxation VAS uses a continuous horizontal line that is 10 centimeters long. On this line, 0 centimeters on the left side represents "unable to relax," while 10 centimeters on the right side represents "extremely relaxed." The closer the mark is to 10 centimeters, the higher the level of relaxation. This scale allows individuals to subjectively indicate their degree of relaxation by marking a point on the line.

CONTACTS AND LOCATIONS:
Overall Officials: Yeu-Hui Chuang, Principal Investigator — Taipei Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Result] Eberhart L, Aust H, Schuster M, Sturm T, Gehling M, Euteneuer F, Rusch D. Preoperative anxiety in adults - a cross-sectional study on specific fears and risk factors. BMC Psychiatry. 2020 Mar 30;20(1):140. doi: 10.1186/s12888-020-02552-w. PMID 32228525
- [Result] Gurler H, Yilmaz M, Turk KE. Preoperative Anxiety Levels in Surgical Patients: A Comparison of Three Different Scale Scores. J Perianesth Nurs. 2022 Feb;37(1):69-74. doi: 10.1016/j.jopan.2021.05.013. Epub 2021 Nov 19. PMID 34810072
- [Result] Gehrig LM. Orthopedic surgery. Am J Surg. 2011 Sep;202(3):364-8. doi: 10.1016/j.amjsurg.2011.06.007. PMID 21871990
- [Result] Greenstein AS, Gorczyca JT. Orthopedic Surgery and the Geriatric Patient. Clin Geriatr Med. 2019 Feb;35(1):65-92. doi: 10.1016/j.cger.2018.08.007. Epub 2018 Oct 11. PMID 30390985
- [Result] Kjaer N, Stabel S, Midttun M. Anti-osteoporotic treatment after hip fracture remains alarmingly low. Dan Med J. 2022 Sep 22;69(10):A01220010. PMID 36205166
- [Result] Konarski W, Pobozy T, Sliwczynski A, Kotela I, Krakowiak J, Hordowicz M, Kotela A. Avascular Necrosis of Femoral Head-Overview and Current State of the Art. Int J Environ Res Public Health. 2022 Jun 15;19(12):7348. doi: 10.3390/ijerph19127348. PMID 35742595
- [Result] Mulugeta H, Ayana M, Sintayehu M, Dessie G, Zewdu T. Preoperative anxiety and associated factors among adult surgical patients in Debre Markos and Felege Hiwot referral hospitals, Northwest Ethiopia. BMC Anesthesiol. 2018 Oct 30;18(1):155. doi: 10.1186/s12871-018-0619-0. PMID 30376809
- [Result] Ruiz Hernandez C, Gomez-Urquiza JL, Pradas-Hernandez L, Vargas Roman K, Suleiman-Martos N, Albendin-Garcia L, Canadas-De la Fuente GA. Effectiveness of nursing interventions for preoperative anxiety in adults: A systematic review with meta-analysis. J Adv Nurs. 2021 Aug;77(8):3274-3285. doi: 10.1111/jan.14827. Epub 2021 Mar 23. PMID 33755246
- [Result] Steghaus S, Poth CH. Assessing momentary relaxation using the Relaxation State Questionnaire (RSQ). Sci Rep. 2022 Sep 29;12(1):16341. doi: 10.1038/s41598-022-20524-w. PMID 36175459
- [Result] Tadesse M, Ahmed S, Regassa T, Girma T, Hailu S, Mohammed A, Mohammed S. Effect of preoperative anxiety on postoperative pain on patients undergoing elective surgery: Prospective cohort study. Ann Med Surg (Lond). 2021 Dec 22;73:103190. doi: 10.1016/j.amsu.2021.103190. eCollection 2022 Jan. PMID 35070278
- [Result] Tulloch I, Rubin JS. Assessment and Management of Preoperative Anxiety. J Voice. 2019 Sep;33(5):691-696. doi: 10.1016/j.jvoice.2018.02.008. Epub 2018 May 9. PMID 29753446
- [Result] Yamamoto K, Nagata S. Physiological and psychological evaluation of the wrapped warm footbath as a complementary nursing therapy to induce relaxation in hospitalized patients with incurable cancer: a pilot study. Cancer Nurs. 2011 May-Jun;34(3):185-92. doi: 10.1097/NCC.0b013e3181fe4d2d. PMID 21252645
- [Result] 譚博謙. (2018). 探討足浴對女大學生焦慮及生理參數之作用. 南華大學自然生物科技學系自然療癒碩士班碩士論文，嘉義縣. 取自 https://hdl.handle.net/11296/gnsfhc